CLINICAL TRIAL: NCT04400266
Title: Buspirone and Melatonin for Depression Following Traumatic Brain Injury
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kaloyan Tanev, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003783
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Depression; Brain Injuries, Traumatic
MeSH Terms: conditions — Depression; Brain Injuries, Traumatic | interventions — Buspirone

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label study of the Buspirone and Melatonin combination administered over 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Buspirone and Melatonin (Experimental): Buspirone 15mg and Melatonin 3mg
  Interventions: Drug: Buspirone; Drug: Mealatonin

INTERVENTIONS:
Drug: Buspirone — Buspirone 15mg once daily
Drug: Mealatonin — Melatonin 3mg once nightly

SUMMARY:
Traumatic brain injuries (TBIs) are common. Post-TBI depression is associated with anxiety, aggression, fatigue, distractibility, anger, irritability, and rumination. The current research group conducted a pilot clinical trial, which investigated the novel treatment combination of buspirone and melatonin (B+MEL) in outpatients with clinical depression. Compared to placebo, B+MEL was associated with a significant improvement in depressive symptoms. Depression following TBI may be different from clinical depression. The B+MEL combination has never been studied in patients with post-TBI depression. The B+MEL has shown promise in ameliorating cognitive difficulties in people with depression. Because cognitive problems are typical in people with post-TBI depression, we plan to measure the effect of the B+MEL combination on cognitive ability in post-TBI depression. Additionally, we are interested in measuring functional magnetic resonance imaging changes before and after treatment with B+MEL in order to gain insight into the brain mechanisms of our hypothesized clinical symptom changes.

The goals of the proposed pilot research project are to assess changes in symptoms in patients with post-TBI depression following Buspirone + Melatonin combination (B+MEL), and the corresponding brain mechanisms underlying these hypothesized changes by measuring: 1) depressive symptoms; 2) cognitive symptoms; 3) functional magnetic resonance imaging.

DETAILED DESCRIPTION:
Background and significance:

Buspirone and Melatonin Combination for the Treatment of Post-TBI Depression Traumatic brain injuries (TBIs) are common (1.7 million cases each year in the US), and major depressive disorder (MDD) occurs in up to 33% of TBI patients. Post- TBI depression is associated with anxiety, aggression, fatigue, distractibility, anger, irritability, and rumination. The current research group conducted a pilot clinical trial, which investigated the novel treatment combination of buspirone (15 mg/day) and melatonin (3mg), in a small outpatient cohort with MDD. Compared to the placebo group, the B+MEL group demonstrated significant improvements in depressive symptoms, at buspirone doses significantly below the recommended therapeutic range for anxiety and recommended dose (40-60 mg) for MDD. Compared to placebo, B+MEL was associated with a significant antidepressant response on the Clinical Global Impressions- Severity (CGI-S, p=0.046) and -Improvement (CGI-I, p=0.04) scales, and on the Inventory of Depressive Symptomatology (IDS, p=0.034). B+MEL was also superior to the pooled buspirone and placebo populations (CGI-S, p=0.009; CGI-I, p=0.021; IDS, p=0.031). This treatment combination has never been studied in patients with post-TBI depression. Depression following TBI may be phenomenologically and neurobiologically distinct from MDD, and the neuroanatomical and biopsychological mechanisms underlying B+MEL response in post-TBI depression are currently unknown. The goal of the proposed pilot research project is to generate pilot data that would serve as a base for an R01 application for a study that will fill this critical gap.

Buspirone and Melatonin Combination and Its Effect on Cognition The current research group compared the effects of B+MEL, buspirone, and placebo on the self-rated Cognitive and Physical Functioning Questionnaire (CPFQ). The CPFQ cognitive dimension score favored the B+MEL combination treatment, compared to the pooled buspirone and placebo groups (p = 0.050). In another randomized, double-blind, SPCD clinical study by the current research group, treatment with NSI-189 - a compound shown to stimulate neurogenesis in in vitro and in vivo, was associated with improvement in cognition, objectively measured by the dimensions of memory (p=0.002) and attention (p=0.048), compared to placebo in MDD patients. The etiology of cognitive impairment in post-TBI depression is complex, and the cognitive changes in response to this novel treatment combination has not been investigated. A possible mechanism of B+MEL action could be the promotion of neurogenesis. Although studying neurogenesis is beyond the scope of the current research, we speculate that a treatment stimulating neurogenesis may contribute to cognitive improvements in post-TBI depression. Hence, we will investigate the effect of B+MEL on cognitive measures of verbal memory, executive functioning, and speed of information processing, in post-TBI depression pre and post-treatment.

Resting State Functional Connectivity in Depression and in TBI MDD is characterized by altered resting state functional connectivity (rsFC) between distinct neural networks. A recent study compared rsFC in TBI with co-morbid depressive symptoms, relative to TBI without depressive symptoms. The results demonstrated increased rsFC between the amygdala and parts of the DAN, salience, somatomotor, and visual networks. Meta-analyses investigating fMRI-based rsFC in MDD demonstrated decreased rsFC within the frontoparietal control network (FPCN), and increased rsFC within the default network (DN). Increased rsFC between the FPCN and DN, and decreased rsFC between the FPCN and dorsal attentional network (DAN) may reflect increased attentional bias toward ruminative thoughts. Decreased rsFC between the affective network (AN) and medial prefrontal cortex may reflect impaired emotional regulation and arousal. Altered rsFC between the ventral attentional network (VAN) and posterior regions may reflect impaired salience detection in MDD. Changes in rsFC have been detected in response to different treatments, such as medication and cognitive behavioral therapy, for depression. Altered rsFC in post-TBI depression is associated with cognitive impairments. A neuroimaging study measuring rsFC in post-TBI depression has not been performed in the context of the novel B+MEL combination treatment. The proposed research is novel with respect to design, technology, and its multi-level integration probing psychological and neurobiological constructs assumed to be critically implicated depression following TBI. Furthermore, it may provide valuable insight regarding rsFC biomarkers implicated in the effective treatment of post-TBI depression.

Specific Aims Specific Aim 1: Assess the changes in depressive symptoms following Buspirone + Melatonin combination (B+MEL) in post-TBI depression.

Hypothesis 1: The B+MEL treatment combination will be associated with improvements in depressive symptoms (changes in HAM-D scores pre- to post-treatment).

Specific Aim 2: Assess the changes in cognitive symptoms following Buspirone + Melatonin combination (B+MEL) in post-TBI depression.

Hypothesis 2: The B+MEL treatment combination will be associated with improvements in measures of verbal memory, executive functioning, and speed of information processing pre- to post-treatment.

Specific Aim 3 (exploratory aim): To assess neuroimaging changes in fMRI resting state functional connectivity in outpatients with post-TBI depression treated with the B+MEL combination.

Hypothesis 3: The B+MEL treatment combination will show pre- to post-treatment resting state functional connectivity increases within the frontoparietal control network (implicated in cognitive control of attention), decreases within the default network (implicated in internally oriented and self-referential thought), and decreases between the frontoparietal control network and the default network.

ELIGIBILITY:
Inclusion Criteria:

Patients with mild or moderate TBI will be included. To be included, a subject must meet the criteria below:

1. Non-penetrating mild or moderate traumatic brain injury that occurred 3 or more months prior to study entry (to minimize natural recovery from TBI)
2. Age: 18-64 years
3. Meeting any one of the following severity criteria, as documented in the patient's medical records:

   1. Glasgow Coma Scale (GCS) score of 9-15 within 4 hours after injury
   2. Loss of consciousness (LOC) >1 minute and <=24 hours
   3. Post-traumatic amnesia (PTA) < 7 days
4. English-speaking
5. Current DSM-5 diagnosis of Major Depressive Episode by medical record diagnosis
6. HAM-D-21 score of 18 or higher
7. Patients who are considered to be appropriate by their clinician and who are willing to be started on Buspirone and Melatonin for clinical purposes.

Exclusion Criteria:

1. History of neurological disorder (e.g., stroke, epilepsy, multiple sclerosis, HIV, neurodegenerative disorders) or any acute or unstable medical condition that is likely to interfere with the assessments or with participation in treatment, as determined by history by the patient or review of their medical records.
2. Evidence from the history of TBI severity greater than moderate, i.e., GCS of 8 or less, LOC > 24 hours, or PTA > 7 days.
3. Inability to attend regular appointments
4. Imminent risk of suicide, as determined by the assessing clinician; HAM-D, Question 3, answers > 1; SDQ, Question 11, answers > 3; spontaneous expressions of suicidal ideation will result in emergency evaluation by a licensed clinician member of study staff for appropriate assessment and triage.
5. Lifetime history of schizophrenia or other primary psychotic disorders, as determined by history by the patient or review of their medical records.
6. History of bipolar disorder, as determined by history by the patient or review of their medical records.
7. Alcohol or substance dependence in the past 3 months, as determined by history by the patient or review of their medical records.
8. Pregnancy or breast-feeding
9. Concomitant use of buspirone, any psychostimulant, or modafinil/armodafinil
10. Patients currently on an antidepressant or who have been on antidepressant in the past 4 weeks
11. Patients with prior intolerances to buspirone or melatonin.
12. Conditions that would preclude a subject from participating in the MRI procedures (e.g., metal implants, aneurysm clips, shrapnel/retained particles, pacemakers, claustrophobia).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Depression | 6 weeks
  Hamilton Depression Rating Scale (HDRS); Min. value: 0; Max, value: 62; Higher number indicates higher severity of symptoms.

SECONDARY OUTCOMES:
Cognition | 6 weeks
  NIH-Toolbox Cognition Battery Fluid Cognition Composite Score

OTHER OUTCOMES:
Functional neuroimaging | 6 weeks
  fMRI resting state functional connectivity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Home Base Program, Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: No